CLINICAL TRIAL: NCT05636332
Title: Philips HeartStart Intrepid 12-lead Electrocardiogram (ECG) Study - The ICE (Intrepid Clinical Engineering) Study
Brief Title: The Intrepid Clinical Engineering Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CCTCECRIntrepid 12Lead2022
Record Dates: First submitted 2022-11-10; First posted 2022-12-05 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Sudden Cardiac Arrest
Keywords: Monitor
MeSH Terms: conditions — Death, Sudden, Cardiac | interventions — Electrocardiography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The qualified electrocardiogram reviewer will be blinded to the age of electrodes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- New electrodes (Other): New package of electrodes
  Interventions: Diagnostic Test: 12 lead Electrocardiogram
- 24-hour opened electrodes (Other): Electrodes opened 24 hours
  Interventions: Diagnostic Test: 12 lead Electrocardiogram
- 30 day opened electrodes (Other): Electrodes opened 30 days
  Interventions: Diagnostic Test: 12 lead Electrocardiogram

INTERVENTIONS:
Diagnostic Test: 12 lead Electrocardiogram — 12 lead Electrocardiogram

SUMMARY:
The purpose of this research study is to collect clinical data to validate a software update for 12-lead electrocardiogram monitoring.

DETAILED DESCRIPTION:
The purpose of this study is to validate the Philips DXL electrocardiogram Algorithm works as intended in the HeartStart Intrepid Monitor/Defibrillator after a software update was completed to address instances of high impedance. This study will also determine the diagnostic quality of the 12-lead electrocardiogram tracing from the HeartStart Intrepid Monitor/Defibrillator.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write, speak, and understand English
* Age: 29 days to 89 years
* Willing and able to provide informed consent and complete study procedures
* Willing to have Philips representatives present during study procedures.

Exclusion Criteria:

* Known allergy to medical adhesives, silicone, or latex (per self-report)
* Any limitation or medical condition, including but not limited to physical or cognitive disability, that would affect the participant's ability to complete study activities (per investigator)
* At the time of enrollment, current enrollment in any other interventional research study
* An employee, or residing family member of an employee, of a company that designs, sells, or manufactures monitor/defibrillator technology or related products (including Philips)

Ages: 29 Days to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El-Gendy, MD, MSc, FCCP, Principal Investigator — Lehigh Pulmonary Associates, PA (D/B/A Florida Lung & Sleep Associates)
Locations (1):
- Lehigh Pulmonary Associates, PA (D/B/A Florida Lung & Sleep Associates), Lehigh Acres, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- New Electrodes: Unopened package of Electrodes will be applied to participants.
- 24-hour Opened Electrodes: Package of Electrodes will be opened 24- hour before applied to participants.
- 30 Day Opened Electrodes.: Package of Electrodes will be opened 30 day (plus or minus 10 days) before applied to participants.
Period: Overall Study
Arm/Group | New Electrodes | 24-hour Opened Electrodes | 30 Day Opened Electrodes.
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Electrodes | 24-hour Opened Electrodes | 30 Day Opened Electrodes | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (18.3) | 31.8 (19.4) | 24.5 (17.0) | 27.0 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 12 | 34
  Male | 10 | 8 | 8 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 12 | 43
  Not Hispanic or Latino | 3 | 6 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Cuban | 3 | 5 | 1 | 9
  Mexican | 9 | 0 | 6 | 15
  Puerto Rican | 0 | 1 | 0 | 1
  White | 7 | 13 | 12 | 32
  Black or African American | 0 | 0 | 1 | 1
  Unknown or not reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Weight [Mean (Standard Deviation); unit: pounds] | 137.2 (65.5) | 160.3 (54.5) | 141.1 (74.6) | 146.2 (65.1)
Height [Mean (Standard Deviation); unit: inches] | 58.7 (14.3) | 61.6 (9.2) | 56.1 (12.1) | 58.8 (12.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (6.1) | 29.4 (8.2) | 29.0 (11.1) | 27.9 (8.8)
Melanin Index [Mean (Standard Deviation); unit: units on a scale] — Melanin index is optical skin parameter related to the melanin content in the tissue. Results are on a broad scale from 0 to 999 over 1 second to detect even the tiniest melanin/redness changes. This measurement is not intended to represent a more favorable tissue condition over other participants in the cohort. The higher the index number, the more pigment is present in the tissue.
  units on a scale | 215.9 (93.6) | 253.8 (96.1) | 226.5 (62.6) | 232.0 (85.5)
Erythema Index [Mean (Standard Deviation); unit: units on a scale] — Erythema Index is optical skin parameter related to the redness content in the tissue. Results are on a broad scale from 0 to 999 over 1 second to detect even the tiniest redness changes. This measurement is not intended to represent a more favorable tissue condition over other participants in the cohort. The higher the index number, the more pigment is present in the tissue.
  units on a scale | 275.8 (94.5) | 316.8 (81.4) | 284.7 (56.0) | 292.4 (79.6)
Skin Temperature [Count of Participants; unit: Participants]
  Hot | 0 | 0 | 0 | 0
  Warm-Normal | 14 | 14 | 13 | 41
  Cool | 6 | 6 | 7 | 19
  Cold | 0 | 0 | 0 | 0
Skin Moisture [Count of Participants; unit: Participants]
  Excessively Dry | 0 | 0 | 0 | 0
  Dry | 20 | 20 | 20 | 60
Skin Texture [Count of Participants; unit: Participants]
  Smooth | 18 | 17 | 19 | 54
  Rough | 0 | 1 | 0 | 1
  Soft | 1 | 0 | 1 | 2
  Firm | 1 | 2 | 0 | 3
Other observations: (Pallor, Jaundiced, Mottled, Cyanotic, etc.) [Count of Participants; unit: Participants] — This measurement was documented as open text for the study team to add any additional skin conditions that were outside of the already described parameters.
  Participants | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Validation of Algorithm Software Update
Description: Number of participants with failure to obtain a 12-lead Electrocardiogram (ECG) with the Philips HeartStart Intrepid Monitor/Defibrillator.
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | New Electrodes | 24-hour Opened Electrodes | 30 Day Opened Electrodes
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

2. Primary Outcome: Diagnostic Quality
Description: Number of participants with diagnostic quality 12-lead ECG tracings from the Philips HeartStart Intrepid Monitor/Defibrillator.
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | New Electrodes | 24-hour Opened Electrodes | 30 Day Opened Electrodes
Number analyzed (Participants) | 20 | 20 | 20
Participants | 20 | 20 | 20

3. Secondary Outcome: Adverse Events
Description: Participants with frequency and severity of unexpected adverse events
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | New Electrodes | 24-hour Opened Electrodes | 30 Day Opened Electrodes
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

4. Secondary Outcome: Unanticipated Adverse Device Effects (UADE)
Description: Participants with unanticipated adverse device effects (UADE).
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | New Electrodes | 24-hour Opened Electrodes | 30 Day Opened Electrodes
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | New Electrodes | 24-hour Opened Electrodes | 30 Day Opened Electrodes
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT05636332/Prot_SAP_000.pdf